CLINICAL TRIAL: NCT02631135
Title: Cognitive Functions After TIVA With Dexmedetomidine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Hale Aksu Erdost, Specialist, Uludag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2007-21/18
Record Dates: First submitted 2015-11-30; First posted 2015-12-16 (Estimated); Results first posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2020-08

CONDITIONS: Postoperative Confusion
Keywords: Dexmedetomidine; cognitive functions; MMSE
MeSH Terms: interventions — Remifentanil; Propofol; Dexmedetomidine; Rocuronium

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1 (TIVA) (Placebo Comparator): Only propofol (started as firstly 12 mg. kg-1 for the 30 minutes, the second 30 minutes 9 mg. kg-1) and remifentanil infusion (0.5 μg.kg-1) and rocuronium for intubation
  Interventions: Drug: Remifentanil; Drug: Propofol; Drug: Rocuronium
- Group 2 (TIVA+D) (Active Comparator): Propofol started as firstly 12 mg. kg-1 for the 30 minutes, the second 30 minutes 9 mg. kg-1) and remifentanil infusion (0.5 μg.kg-1),and also dexmedetomidine infusion (started as 0.5 μg.kg-1 without making the loading dose and the dose change was not made during the operation) and rocuronium for intubation
  Interventions: Drug: Remifentanil; Drug: Propofol; Drug: Dexmedetomidine; Drug: Rocuronium

INTERVENTIONS:
Drug: Remifentanil — In case of tachycardia or hypertension the opioid dose was reduced, in case of bradycardia or hypertension the opioid dose was increased
  Other Names: ultiva
Drug: Propofol — BIS values were arranged 40-60 until the end of operation
Drug: Dexmedetomidine — 0.5 microgram/kg infusion, no changes
  Other Names: precedex
  Arms: Group 2 (TIVA+D)
Drug: Rocuronium — 0.5 mg/kg iv for intubation, no changes
  Other Names: esmeron

SUMMARY:
It is important to wake up without any problem and comfortably from the general anesthesia. The aim of this study is to investigate the effects of addition dexmedetomidine to the balanced intravenous anesthesia with propofol over the cognitive functions and also it is considered that the addition of dexmedetomidine would reduce the use of anesthetics drugs in TİVA. Together with this effects, it has been considered that the disorder of the cognitive functions in postoperative period and the need for anesthetic drugs in postoperative period will be less.

After the approval of the Ethics Committee and the patients being informed and taking informed consent from them 18 female 23 male totally 41 patients between the age of 20-60 years old, who had lumbar disc hernia, under general anesthesia have been taken under the study. The patients have been divided into two groups by closed envelope drawing method, randomly. All patients cognitive functions were evaluated by MMSE (Mini Mental State Examination) during the premedication visit. For this study group Standardized Mini Mental Test Examination (SMMT-E) were used, which has quite practical usage, for the untrained patients, and test composed of question-answer in order to calculate the remembering, caution and calculation structure and the scores were recorded. All patients had received the same anesthesia induction with propofol infusion (started at firstly 12 mg. kg-1 for the 30 minutes, the second 30 minutes 9 mg. kg-1 and the BIS(bispectral index) values were arranged between 40-60 until the end of the operation), and remifentanil infusion (0.5 μg.kg-1 was applied as opioid and was arranged according to the tension artery and heart rate). In the dexmedetomidine group, dexmedetomidine infusion had started as 0.5 μg.kg-1 without making the loading dose and the dose change was not made. Rocuronium 0.5 mg. kg-1 iv. was applied for the endotracheal intubation. After the operation all patients have taken to the recovery room.

Then the tests of cognitive function evaluation were repeated as postoperative 2nd hour, 24 hours, 1 week and 1 month.

DETAILED DESCRIPTION:
After the approve of the Ethics Committee and the patients were informed and taken informed consent form from them (18 female and 23 male) totally 41 patients between the age of 20-60 years old, who had lumbar disc hernia, under general anesthesia have been taken under the study. The patients with hepatic, renal or neurological diseases and using sedative- hypnotic, anticonvulsive and stimulant drugs and pregnant patients were excluded. Then they have been divided into two groups by closed envelope drawing method randomly and were allowed to stay hungry at least 8 hours. All the patients were applied the cognitive functions during the premedication visit MMSE (Mini Mental State Examination) that has quite practical usage and the test called Standardized Mini Mental Test Examination(SMMT-E) for the untrained persons. Test composed of question-answer in order to calculate the remembering, caution and calculation structure. All patients SMMTE scores were recorded. In the operation room, patients were applied the standard D-II derivation electrocardiography, heart beat rate, non-invasive arterial pressure, peripheral oxygen saturation (SpO2) and Bispectral Index (BİS) monitorization. Serum sale infusion was started by opening the vascular access with 18-20 gauge cannula. The skin of forehead and the temporal side were cleaned with alcohol cotton for the BİS monitorization. The electrode in the proximal part of the three electrodes of disposable BİS sensor was adhered to the middle of the forehead; the distal electrode to the temporal area on the eye line and the other electrode in between them both were adhered. The BİS values (BİS Monitor, Aspect, USA) were continuously monitored. The Group I (TİVA, n= 20) were received propofol-remifentanil and the Grup II (TİVA+D, n= 20) propofol- remifentanil and additional dexmedetomidine infusion.

Induction of propofol infusion in all two groups was started as firstly 12 mg. kg-1 for the 30 minutes, the second 30 minutes 9 mg. kg-1 and the BIS values were arranged between 40-60 until the end of the operation. At the same time remifentanil infusion 0.5 μg.kg-1 was applied as opioid and arranged according to the tension artery and heart rate. The dexmedetomidine infusion has been started as 0.5 μg.kg-1 without making the loading dose and the dose change was not made. Rocuronium 0.5 mg. kg-1 iv. was applied for the endotracheal intubation. After intubation the carbon dioxide concentration was recorded in all periods.

The patients were ventilated mechanically after the intubation in order to be ETCO2 (end-tidal carbon dioxide) 30-44 mmHg, tidal volume 8-10 mL. kg-1 . In case of tachycardia or hypertension the opioid dose was reduced in case of bradycardia or hypertension while the opioid dose was being increased. Propofol infusion was arranged to be kept in between BİS score 40-50. The effect of the used muscle relaxant was returned by neostigmine 0,05- 0,07 mg. kg-1 i.v. and atropin 0,03 mg. kg -1 i.v. After the operation all patients have been taken to the recovery room.

Then the tests of cognitive function evaluation were repeated as postoperative 2nd hour, 24 hours, 1 week and 1 month.

ELIGIBILITY:
Inclusion Criteria:

* under going lumbar disk hernia operation
* 20-60 years old
* ASA (American Society of Anesthesiologists Physical Status classification) classification I-II

Exclusion Criteria:

* pregnants
* Patients with hepatic, renal or neurological diseases and
* patients using sedative- hypnotic, anticonvulsive and stimulant drugs
* One of the patient excluded from the study (can not be able to reached after surgery)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-01; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hulya Bilgin, professor, Study Director — Uludag University
Locations (1):
- Uludag University, Bursa, Turkey (Türkiye)

REFERENCES:
- [Background] Molloy DW, Standish TI. A guide to the standardized Mini-Mental State Examination. Int Psychogeriatr. 1997;9 Suppl 1:87-94; discussion 143-50. doi: 10.1017/s1041610297004754. PMID 9447431
- [Background] Magni G, Baisi F, La Rosa I, Imperiale C, Fabbrini V, Pennacchiotti ML, Rosa G. No difference in emergence time and early cognitive function between sevoflurane-fentanyl and propofol-remifentanil in patients undergoing craniotomy for supratentorial intracranial surgery. J Neurosurg Anesthesiol. 2005 Jul;17(3):134-8. doi: 10.1097/01.ana.0000167447.33969.16. PMID 16037733
- [Background] Gurbet A, Basagan-Mogol E, Turker G, Ugun F, Kaya FN, Ozcan B. Intraoperative infusion of dexmedetomidine reduces perioperative analgesic requirements. Can J Anaesth. 2006 Jul;53(7):646-52. doi: 10.1007/BF03021622. PMID 16803911
- [Result] Weinbroum AA, Geller E. Flumazenil improves cognitive and neuromotor emergence and attenuates shivering after halothane-, enflurane- and isoflurane-based anesthesia. Can J Anaesth. 2001 Nov;48(10):963-72. doi: 10.1007/BF03016585. PMID 11698314
- [Result] Kostopanagiotou G, Markantonis SL, Polydorou M, Pandazi A, Kottis G. Recovery and cognitive function after fentanyl or remifentanil administration for carotid endarterectomy. J Clin Anesth. 2005 Feb;17(1):16-20. doi: 10.1016/j.jclinane.2004.03.008. PMID 15721724

RESULTS

PARTICIPANT FLOW:
Recruitment Details: patients, who scheduled to have general anesthesia for surgery of a prolapsed lumbar disc
Pre-assignment Details: pregnant patients and those with hepatic, renal or neurological disease and those using sedative, hypnotic, anticonvulsive or stimulant drugs were excluded from the trail before assignment to groups and one patient excluded from the study (can not be able to reach after surgery)
Groups:
- Group 1 (TIVA): Only propofol (started as firstly 12 mg. kg-1 for the 30 minutes, the second 30 minutes 9 mg. kg-1) and remifentanil infusion (0.5 μg.kg-1)
  Remifentanil: In case of tachycardia or hypertension the opioid dose was reduced, in case of bradycardia or hypertension the opioid dose was increased
  Propofol: BIS (bispectral index) values were arranged 40-60 until the end of operation
  Rocuronium: 0.5 mg/kg iv for intubation, no change
- Group 2 (TIVA+D): Propofol started as firstly 12 mg. kg-1 for the 30 minutes, the second 30 minutes 9 mg. kg-1) and remifentanil infusion (0.5 μg.kg-1),and also dexmedetomidine infusion (started as 0.5 μg.kg-1 without making the loading dose and the dose change was not made during the operation)
  Remifentanil: In case of tachycardia or hypertension the opioid dose was reduced, in case of bradycardia or hypertension the opioid dose was increased
  Propofol: BIS values were arranged 40-60 until the end of operation
  Dexmedetomidine: 0.5 microgram/kg infusion, no changes
  Rocuronium: 0.5 mg/kg iv for intubation, no change
Period: Overall Study
Arm/Group | Group 1 (TIVA) | Group 2 (TIVA+D)
Started | 21 | 20
Completed | 20 | 20
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1 (TIVA): Only propofol (started as firstly 12 mg. kg-1 for the 30 minutes, the second 30 minutes 9 mg. kg-1) and remifentanil infusion (0.5 μg.kg-1)
  Remifentanil: In case of tachycardia or hypertension the opioid dose was reduced, in case of bradycardia or hypertension the opioid dose was increased
  Propofol: BIS values were arranged 40-60 until the end of operation
  Rocuronium: 0.5 mg/kg iv for intubation, no change
- Total: Total of all reporting groups
Arm/Group | Group 1 (TIVA) | Group 2 (TIVA+D) | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.60 (11.5) | 41.65 (10.1) | 43.62 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 11 | 12 | 23
Region of Enrollment [Number; unit: participants]
  Turkey | 21 | 20 | 41
weight [Mean (Standard Deviation); unit: kg] | 75.7 (8.8) | 84.1 (13.1) | 79.9 (11.83)
height [Mean (Standard Deviation); unit: cm] | 168.65 (7.84) | 173.4 (10.2) | 171.02 (9.31)
Mini Mental State examination [Mean (Full Range); unit: units on a scale] — The Total score range of MMSE is 0-30, and the higher score indicates better cognitive function.
  units on a scale | 29.15 [24 to 30] | 28.60 [26 to 30] | 28.87 [24 to 30]

OUTCOME MEASURES:

1. Primary Outcome: Mini Mental State Examination (MMSE) Score at the Second Hour After Surgery
Description: The cognitive function evaluation performed by MMSE test at the second hour of the surgery The Total score range of MMSE is 0-30, and the higher score indicates better cognitive functions
Time Frame: Postoperative hour 2
Population: per protocol
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Group 1 (TIVA) | Group 2 (TIVA+D)
Number analyzed (Participants) | 21 | 20
scores on a scale | 27.40 (1.31) | 26.45 (1.19)

2. Primary Outcome: Mini Mental State Examination (MMSE) Score at the First Month After Surgery
Description: The cognitive function evaluation performed by MMSE test at the one month of the surgery The Total score range of MMSE is 0-30, and the higher score indicates better cognitive functions
Time Frame: Postoperative month one
Population: per protocol
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Group 1 (TIVA) | Group 2 (TIVA+D)
Number analyzed (Participants) | 20 | 20
scores on a scale | 29.15 (1.18) | 28.65 (1.08)

3. Primary Outcome: Mini Mental State Examination (MMSE) Score at the First Week After Surgery
Description: The cognitive function evaluation performed by MMSE test at the one week of the surgery The Total score range of MMSE is 0-30, and the higher score indicates better cognitive functions
Time Frame: postoperative week one
Population: per protocol
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Group 1 (TIVA) | Group 2 (TIVA+D)
Number analyzed (Participants) | 20 | 20
scores on a scale | 28.95 (1.31) | 28.15 (1.26)

4. Primary Outcome: Mini Mental State Examination (MMSE) Score at the 24th Hour After Surgery
Description: The cognitive function evaluation performed by MMSE test at the 24th hour of the surgery The Total score range of MMSE is 0-30, and the higher score indicates better cognitive functions
Time Frame: Postoperative hour 24
Population: per protocol
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Group 1 (TIVA) | Group 2 (TIVA+D)
Number analyzed (Participants) | 21 | 20
scores on a scale | 29.05 (1.23) | 28.60 (1.09)

ADVERSE EVENTS:
Time Frame: 1 month
Description: questionnaire postoperative 2, 12, 24 hour and after 1 month
Arm/Group | Group 1 (TIVA) | Group 2 (TIVA+D)
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
The examined subject number was small The evaluation of cognitive function was made by one test which is very associate with the participants education level

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No